CLINICAL TRIAL: NCT02964481
Title: Donation of Blood for Genetic Testing With Clinical Data From the North American Malignant Hyperthermia Registry
Brief Title: Malignant Hyperthermia Registry and Genetic Testing
Status: Terminated | Type: Observational
Why Stopped: Lack of funding to enroll additional participants
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-1749
Record Dates: First submitted 2016-06-29; First posted 2016-11-16 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Malignant Hyperthermia
Keywords: malignant; genetics; RYR1; CAC-NA1S; hyperthermia
MeSH Terms: conditions — Malignant Hyperthermia; Hyperthermia | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be used to extract DNA for genotyping, pyrosequencing and pluripotent stem cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Malignant Hyperthermia Phenotype cases: Samples from persons who identify as having the malignant hyperthermia phenotype by the North American MH Registry (NAMHR)
  Interventions: Genetic: Whole exome sequencing
- Caffeine Halothane Contracture Test negative controls: Controls who had negative Caffeine Halothane Contracture Test (CHCT) from North American MH Registry (NAMHR)
  Interventions: Genetic: Whole exome sequencing

INTERVENTIONS:
Genetic: Whole exome sequencing — DNA sequencing of protein coding sections of all genes

SUMMARY:
The purpose of this study is to to determine the penetrance of known and probable pathogenic variants in genes and the factors that contribute to penetrance in a population of children and adults in the United States exposed to Malignant Hyperthermia (MH) trigger agents.

DETAILED DESCRIPTION:
The purpose of the study is to determine how genetic mutations and variants in combination with non-genetic factors influence risk for MH in children who had general anesthesia with triggering agents and develop reliable predictive MH risk algorithms. Rationale: Once the factors responsible for MH risk are determined, it will be possible to better predict risk and develop better individualization of anesthetics such as tailored selection of intravenous anesthetics, regional anesthesia and avoidance of all triggering agents. The long-term goal is to tailor and improve safety of anesthetic and clinical care and to reduce mortality, morbidity and cost of care due to MH with right anesthetics and muscle relaxants for endotracheal intubations for an individual child.

ELIGIBILITY:
Inclusion Criteria:

* Any English speaking person registered at NAHMR who has had a positive clinical manifestation of Malignant Hyperthermia
* Any person with a positive Caffeine Halothane Contracture probTest (CHCT) or a close relative of a person that had these.

Exclusion Criteria:

* Any person who has NOT had a positive clinical manifestation of Malignant Hyperthermia
* Any person with a positive Caffeine Halothane Contracture Test (CHCT) or NOT a close relative of a person that had these. Non-English speaking registrants will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with documented MH clinical presentation and CHCT negative controls from NAMHR
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Genetic comparison of MH phenotype subjects to that of the CHCT negative control subjects. | Within data collection period (5 years total).
  MHS subjects and CHCT negative controls recruited from the North American MH Registry will have whole genome sequencing

SECONDARY OUTCOMES:
Genomic factors that influence Malignant Hyperthermia. | Within data collection period (5 years total).
  A Batesian inference algorithm based on multiple genetic risk factors assessed from DNA data collected
Induced pluripotent stem cells will be used for functional testing and gene editing | Indefinite - dependent on funding
  Induced pluripotent stem cells will be made for future in-vitro analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Sadhasivam S, Brandom BW, Henker RA, McAuliffe JJ. Bayesian modeling to predict malignant hyperthermia susceptibility and pathogenicity of RYR1, CACNA1S and STAC3 variants. Pharmacogenomics. 2019 Sep;20(14):989-1003. doi: 10.2217/pgs-2019-0055. PMID 31559918